CLINICAL TRIAL: NCT01714713
Title: A Multicenter 26-Week Extension Study to Evaluate the Safety and Clinical Effects of Prolonged Exposure to Two Doses of EVP-6124, an Alpha-7 Nicotinic Acetylcholine Receptor Agonist, as an Adjunctive Pro-cognitive Treatment in Subjects With Schizophrenia on Chronic Stable Atypical Antipsychotic Therapy
Brief Title: A 26-Week Extension Study of EVP-6124 (Alpha-7 nAChR) as an Adjunctive Pro-Cognitive Treatment in Schizophrenia Subjects on Chronic Stable Atypical Antipsychotic Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: FORUM Pharmaceuticals Inc (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EVP-6124-017; 2012-003228-19 (EudraCT Number)
Record Dates: First submitted 2012-10-19; First posted 2012-10-26 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2015-09

CONDITIONS: Schizophrenia; Impaired Cognition
Keywords: Schizophrenia; Cognition; Cognition Impairment; Alpha-7 nAChR
MeSH Terms: conditions — Schizophrenia; Cognition Disorders | interventions — 7-chloro-N-quinuclidin-3-yl-benzo(b)thiophene-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EVP-6124 low dose (Experimental): low dose Tablet, Once Daily, Day 1 through Day 182
  Interventions: Drug: EVP-6124
- EVP-6124, high dose (Experimental): high dose Tablet, Once Daily, Day 1 through Day 182
  Interventions: Drug: EVP-6124

INTERVENTIONS:
Drug: EVP-6124 — Arm 1, 2

SUMMARY:
This study is being conducted to further investigate the safety of prolonged exposure to EVP-6124 in subjects with Schizophrenia receiving a stable dose of an atypical antipsychotic who completed double-blind treatment on studies EVP-6124-015 and EVP-6124-016.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the Day 182 visit in a previous 26-week double-blind study (EVP-6124-015 or EVP-6124-016).
* Subject has signed informed consent for this extension study, indicating that the subject understands the purpose of and procedures required for the study, before the initiation of any extension study specific procedures. Subjects who are unable to provide informed consent will not be included in the study
* No clinically significant changes in the subject's medical status during the participation in EVP-6124-015 or EVP-6124-016. Any significant changes in health care status and their impact on subject eligibility will be reviewed by the investigator and sponsor on a case-by-case basis.
* In the opinion of the investigator, the extension treatment is in the best interest of the subject.
* Fertile, sexually active subjects (men and women) must use an effective method of contraception during the study. Females and the female partners of male must be surgically sterile (hysterectomy or bilateral tubal ligation), postmenopausal for at least 1 year, willing to practice adequate methods of contraception if of childbearing potential (defined as consistent use of combined effective methods of contraception [including at least one barrier method]). Female subjects must have a negative urine pregnancy test predose on Day 1.

Exclusion Criteria:

* Significant risk for suicidal or violent behavior, as determined by the investigator. Significant risk for suicidal behavior is defined as 1) suicidal ideation as endorsed on items 4 and 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS); 2) suicidal behaviors detected by the C-SSRS; or 3) psychiatric interview and examination.
* Adverse events from the previous study (EVP-6124-015 or EVP-6124-016) that have not resolved, are of moderate or greater severity and judged to be possibly related or related to study drug and are thought by the investigator to be contraindications to study participation.
* Any condition which would make the subject, in the opinion of the investigator, unsuitable for the study.
* Female subjects who are pregnant.
* Subjects who received any other investigational treatment during participation in either EVP-6124-015 or EVP-6124-016 other than assigned study medication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 830 (Actual)
Dates: Start 2013-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of EVP-6124 or Placebo in Subjects with Schizophrenia | Baseline through Day 182 or Early Termination
  All adverse experiences spontaneously reported by subject and/or observed by investigator and repeated clinical evaluation of physical examinations, vital signs, 12-lead ECG (electrocardiogram), ambulatory ECG, and laboratory tests (hematology/blood/chemistry/urinalysis)

SECONDARY OUTCOMES:
Change from Baseline in the Clinical Global Impression (CGI) - Severity (CGI-S) to Day 182 | Baseline to Day 182 or Early Termination
Change from Baseline in the Clinical Global Impression (CGI) - Change (CGI-C) to Day 182 | Baseline to Day 182 or Early Termination
Change from Baseline in the EuroQol-5D (EQ-5D-5L) to Day 182 | Baseline to Day 182 or Early Termination
Change from Baseline in the Columbia Suicide Severity Rating Scale (C-SSRS) to Day 182 | Baseline to Day 182 or Early Termination
Change from Baseline in the Client Socio-Demographic and Service Receipt Inventory-European Version (CSSRI-EU) to Day 182 | Baseline to Day 182 or Early Termination

CONTACTS AND LOCATIONS:
Locations (128):
- United States (69):
  - Little Rock, Arkansas
  - Anaheim, California
  - Bellflower, California
  - Cerritos, California
  - Chino, California
  - Costa Mesa, California
  - Culver City, California
  - Downey, California
  - Escondido, California
  - Garden Grove, California
  - Glendale, California
  - Los Angeles, California
  - Mesa, California
  - Norwalk, California
  - Oakland, California
  - Oceanside, California
  - Orange, California
  - Riverside, California
  - San Diego, California
  - San Gabriel, California
  - Santa Ana, California
  - Sherman Oaks, California
  - Torrance, California
  - Washington D.C., District of Columbia
  - Lauderhill, Florida
  - Miami, Florida
  - Miami Springs, Florida
  - North Miami, Florida
  - Oakland Park, Florida
  - Orange City, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Smyrna, Georgia
  - Chicago, Illinois
  - Oak Brook, Illinois
  - Oak Park, Illinois
  - Wichita, Kansas
  - Lake Charles, Louisiana
  - Shreveport, Louisiana
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Flowood, Mississippi
  - Creve Coeur, Missouri
  - O'Fallon, Missouri
  - Saint Charles, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Nashua, New Hampshire
  - Princeton, New Jersey
  - Albuquerque, New Mexico
  - Cedarhurst, New York
  - Jamaica, New York
  - New York, New York
  - Charlotte, North Carolina
  - Cleveland, Ohio
  - Shaker Hts., Ohio
  - Oklahoma City, Oklahoma
  - Conshohocken, Pennsylvania
  - Jenkintown, Pennsylvania
  - Norristown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Phoenixville, Pennsylvania
  - Austin, Texas
  - Dallas, Texas
  - Salt Lake City, Utah
  - Bellevue, Washington
  - Spokane, Washington
- Argentina (3):
  - La Plata, Buenos Aires
  - Mendoza, Mendoza Province
  - C.a.b.a
- Australia (2):
  - Adelaide, South Australia
  - Melbourne, Victoria
- Mechelen, Belgium
- Canada (5):
  - Calgary, Alberta
  - Penticton, British Columbia
  - Chatham, Ontario
  - Kingston, Ontario
  - Montreal, Quebec
- Colombia (5):
  - Medellín, Antioquia
  - Barranquilla, Atlántico
  - Pereira, Risaralda Department
  - Bogota D.C.
  - Bogota D.C
- Germany (5):
  - Berlin
  - Düsseldorf
  - Leipzig
  - Mittweida
  - Stralsund
- Italy (3):
  - Catania, CT
  - Milan, Milano
  - Roma, RM
- Mexico (5):
  - Guadalajara, Jalisco
  - Mexico City, Mexico City
  - Monterrey, Nuevo León
  - San Luis Potosí City, San Luis Potosí
  - Mexico City
- Bełchatów, Poland
- Romania (7):
  - Campulung Muscel, Argeş
  - Oradea, Bihor County
  - Cluj-Napacu, Cluj
  - Cluj-Napoca, Cluj
  - Palazu Mare, Constanța County
  - Târgu Mureş, Mureș County
  - Bucharest, Sector 4
- Russia (6):
  - Talagi, Arkhangelskaya oblast
  - Smolensk, Smolensk Oblast
  - Moscow
  - Saint Petersburg
  - Stavropol
  - Yaroslavl
- Singapore, Singapore, Singapore
- Spain (5):
  - Salamanca, Castille and León
  - Zamora, Castille and León
  - Alcorcón, Madrid
  - Coslada, Madrid
  - Madrid, Madrid
- Ukraine (9):
  - Vil. Stepanivka, Kherson Oblast
  - Dnipropetrovsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kyiv
  - Lviv
  - Poltara
  - Poltava
  - Vinnytsia
- London, United Kingdom